CLINICAL TRIAL: NCT04514055
Title: Evaluation of a De-epithelialized Free Gingival Connective Tissue Graft Wall Technique in Management of Cairo's RT2 and RT3 With Intra-bony Defects: A Case Series
Brief Title: Connective Tissue Graft Wall Technique in Management of Cairo's RT2 and RT3 With Intra-bony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Galal Bendary, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14422019493595
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Recession, Gingival
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- De-epithelialized connective tissue graft wall (Experimental): Simplified papilla preservation flap will be applied in the narrow interproximal spaces (≤2 mm), where an oblique incision starting from the gingival margin at the buccal-line angle of the involved tooth reaching the mid-interproximal portion of the papilla under the contact point of the adjacent tooth will be performed using a 15c blade.
  A free gingival graft will be obtained from the hard palate and de-epithelized extra-orally.
  A Coronally advanced flap will be performed. The de-epithelialized FGG will be sutured coronally using a 6-0 vicryl suture to the anatomical papillae of the two teeth adjacent to the defect and apically to the periosteum left in place apical to the exposed bone.
  The flap will be sutured using internal Horizontal mattress suture at the base of the simplified papilla and a vertical mattress suture will be placed in a more coronal position so complete soft tissue closure can be obtained.
  Interventions: Procedure: De-epithelialized connective tissue graft wall

INTERVENTIONS:
Procedure: De-epithelialized connective tissue graft wall — A de-epithelialized free gingival connective tissue graft will be used to treat Cairo's recession type 2 and type 3 associated with inta-bony defects

SUMMARY:
Recession presents a day to day challenge due to the high esthetic demand of the patients. The prevalence, extent, and severity of recession associated with intra-bony defects due to periodontitis increases with age rendering the success of the root coverage procedures questionable due to loss of interdental papillary support. .

Therefore, connective tissue graft wall technique in cases of Cairo's RT2 and RT3 gingival recession associated with intra bony defects seems promising with regard to recession depth reduction and radiographic bone fill.

DETAILED DESCRIPTION:
Recession is usually treated by an array of mucogingival surgical techniques. The choice of the procedure depends on the morphology of the recession defect. Full root coverage in RT2 and RT3 gingival recession defects cannot always be predictably achieved due to the presence of bone loss. Improvement is further complicated when these recessions are associated with intra-bony defects as mucogingival surgical techniques are not designed to treat intra-bony defects. The preferred surgical modality for treatment of intrabony defects is guided tissue regeneration. However when considering recession defects, the amount of root coverage achieved by GTR may be limited with less results achieved.

Most of the root coverage procedures have proven to be successful, however, when recession is associated with intrabony defect especially in cases of low height and thickness of keratinized tissue and GTR is performed, the treatment results were unpredictable and it was found that the recession might increase post-surgically, so the procedure might offer a limited benefit.

Therefore, the technique introduced by Zucchelli et al. in 2014 in cases of RT2 and RT3 gingival recession associated with intra bony defects seems promising with regard to recession depth reduction and radiographic bone fill. A simplified papilla preservation technique was performed on the defect site, a de-epithelialized free gingival graft was used to treat the gingival recession present and intrabony defects because it acted as a membrane, creating a buccal wall to the intra-bony defect from one side and on the palatal aspect since no flap elevation was done. The palatal connective tissue acted as a palatal wall preventing gingival epithelium and connective tissue from contacting the space created allowing both improved root coverage and bone fill. He reported interproximal probing depth reduction, clinical attachment gain, improvement in the papilla covering the intrabony defect regarding the gingival thickness and root coverage and complete bone fill was shown radiographically in 1 year.

This technique needs more investigations, but it seems encouraging to improve regenerative and esthetic parameters in the treatment of deep infrabony defects, in one surgical session.

ELIGIBILITY:
Inclusion Criteria:

* Teeth with buccal RT2 and RT3 recession associated with an intra-bony defect on single rooted teeth.
* Single and multiple recessions.
* Full mouth plaque score (FMPS )<20% at baseline.
* Full mouth bleeding score (FMBS )<10% at baseline.
* Systemically healthy.
* Cooperative patients.

Exclusion Criteria:

* Smokers.
* Pregnancy and lactation.
* Stage 4 Grade C periodontitis.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Gingival recession depth | Changes at 3 and 6 months post-operative
  Measured from the cementoenamel junction to the gingival margin using a William's graduated periodontal probe. The probe will be inserted into the sulcus gently parallel to the long axis of the tooth.

SECONDARY OUTCOMES:
Radiographic bone fill | At 6 months post-operative
  The depth of intra-bony defect (IBD) will be measured from the alveolar bone crest to the base of the defect at baseline and after six months to detect the amount of bone fill. Individually customized bite blocks will be created for the patients using alginate impression material and acrylic resin. Parallel-angle technique will be used to obtain standardized radiographs
Gingival Recession Width | Changes at 3 and 6 months post-operative
  Horizontal distance will be measured from one border of the recession to another in mesio-distal direction at CEJ level
Percentage of Root Coverage | Changes at 3 and 6 months post-operative
  Percentage of root coverage will be calculated by obtaining the baseline recession depth, postoperative recession depth and will be calculated according to the following formula:
  (Baseline RD-6 months RD)/(Baseline RD) ×100
Gingival Thickness | Changes at 3 and 6 months post-operative
  Measured 2 mm apical to the gingival margin with a short needle for and a 3 mm diameter silicon disk stop. The needle is inserted perpendicular to the mucosal surface, through the soft tissues with light pressure until resistance is found due to presence of bone. The silicone disc stop on the spreader was placed in tight contact with the external gingival tissue surface. After carefully removing the spreader, penetration depth was measured with William's periodontal probe
Probing Depth | Changes at 3 and 6 months post-operative
  Measured from the gingival margin to the bottom of the gingival sulcus using William's periodontal probe with the probe inserted parallel to the long axis of the tooth
Clinical Attachment Level | At 3 and 6 months post-operative
  Measured from the CEJ to the bottom of the gingival sulcus using William's periodontal probe.
Width of the Keratinized Tissue | At 3 and 6 months post-operative
  Measured from the gingival margin to the muco-gingival junction using William's periodontal probe.
Post-Operative Pain | At 7 and 14 days post-operative
  Visual Analogue Scale (VAS) with numbers from 0 to 10 ('no pain' to 'the most painful) measured daily for the first 2 weeks postoperatively
Post-Operative patient's Satisfaction | At 6 months post-operative
  A 3-item questionnaire is asked and the patients shall use a 7-point answer scale
Bleeding on Probing | At 6 months post-operative
  BOP score will be assessed as the number of bleeding sites (dichotomous yes/no evaluation) when stimulated by a standardized periodontal probe with a controlled (∼25 g) force to the bottom of the sulcus at six sites (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, disto-lingual) on all present teeth
Plaque Index | At 6 months post-operative
  PI will be assessed using a standardized periodontal probe to agitate the gingival margin and assessing the presence or absence of plaque at the margin. This will be recorded at 4 sites per tooth on all teeth

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Bendary, Principal Investigator — Cairo University
Locations (1):
- Faculty of dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol, informed consent, clinical study report
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After completion of the study
Access Criteria: ClinicalTrials.gov
URL: http://ClinicalTrials.gov